CLINICAL TRIAL: NCT01548300
Title: Environmental Triggers Of Cardiometabolic Disease
Acronym: AIRCMD
Status: Completed | Type: Observational
Sponsor: Sanjay Rajagopalan (Other)
Collaborators: University of Michigan (Other); Peking Union Medical College (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor-Investigator, Sanjay Rajagopalan, Professor, University of Maryland
Organization: University of Maryland, Baltimore (Other)
Other Study IDs: HP-00059994; R01ES019616 (NIH)
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Metabolic Syndrome X
Keywords: cardiometabolic disease
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enrolled participants: Subjects will be recruited from clinics affiliated with the Fuwai Hospital, PUMC. The participants will be nonsmokers with cardiometabolic disease, that are not taking anti-hypertensive, glucose-lowering, or lipid-lowering medications or drugs that alter baseline insulin sensitivity, blood pressure, or endothelial function, daily use of NSAIDS is not allowed.

SUMMARY:
The investigators posit that a multi-national collaborative effort with focused investigations in environments with the highest levels of exposure (developing countries such as China and India), are likely to provide new and much needed data on the risk posed by these variables on an individuals life-time risk for type 2 diabetes and cardiovascular complications. The investigators will test this hypothesis through the establishment of a network that would lead studies on the links between exposure and adverse Chronic cardiometabolic effects and propose doing this in this as part of 3 specific aims.

DETAILED DESCRIPTION:
In aim 1, the investigators propose to establish feasibility of such an effort in Beijing, China, an effort that will involve implementation of novel exposure assessment methodologies simultaneously with the ability to execute key surrogate outcome measures of importance in cardiovascular risk with CM diseases. In Aim 2, the association between functional cardiovascular risk variables [insulin sensitivity, Blood Pressure, endothelial function] and acute and sub-acute variations in personal black carbon and ambient particulate matter 2.5 levels among 50 individuals with the chronic cardiometabolic syndrome will be investigated. In Aim 3, the investigators will examine potential biologic pathways of importance in the proposed functional outcomes. Specifically the investigators will determine the association between ambient particulate matter 2.5 levels and alterations in adipocytokines/inflammatory variables and autonomic nervous system balance.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmokers, 35-65 years living in a nonsmoking household.
* CM will be defined by IDF criteria (http://www.idf.org) specific for Asians [waist circumference >90 cm in males and 80 cm in females) plus any two of the following four factors: TG level: >150 mg/dL, HDL: < 40 mg/dL in males and < 50 mg/dL in females, systolic BP >130, fasting plasma glucose > 100 mg/dL or previously diagnosed type 2 diabetes.

Exclusion Criteria:

* Any active smoking within past 1 year, occupational exposures to pollutants (per discretion of investigators), self-reported daily secondhand smoke exposure > 1 hour long (workplace or home),
* History of any CV disease (e.g. previous myocardial infarction), or overt type 2 diabetes.
* Fasting glucose > 126 mg/dL or a screening BP is >160/100 mm Hg.
* Patients cannot be taking any anti-hypertensive, glucose-lowering, or lipid-lowering medications or drugs that can alter baseline insulin sensitivity, BP, or endothelial function (e.g. anti-oxidants, multi-vitamins, folic acid, fish oil supplementation, L-arginine),
* Daily use of NSAIDS is not allowed; however intermittent PRN usage is acceptable.

In the course of the year should a subject develop any of exclusion criteria they will be allowed to complete the study and the potential confounding effects will be assessed in statistical analyses.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from clinics affiliated with the Fuwai Hospital, PUMC. The participants will be nonsmokers with cardiometabolic disease, that are not taking anti-hypertensive, glucose-lowering, or lipid-lowering medications or drugs that alter baseline insulin sensitivity, blood pressure, or endothelial function, daily use of NSAIDS is not allowed.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Death | 48 months
  Death, MI (fatal and non-fatal), target vessel revascularization and hospitalization for angina at 6 months

SECONDARY OUTCOMES:
Inflammation markers | 30 days
  EPC counts and measurement of LyC6hi, CD11b+ cells

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Rajagopalan, MD, Principal Investigator — Ohio State University; Dongfeng GU, MD, Principal Investigator — Peking Union Medical College; Brook Robert, MD, Principal Investigator — University of Michigan
Locations (3):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - The Ohio State University, Columbus, Ohio
- Peking Union Medical College, Beijing, Beijing Municipality, China